CLINICAL TRIAL: NCT01535456
Title: A Pilot Study for Using 18F-FLT PET Imaging To Assess Response In Patients With Myelodysplastic Syndrome (MDS) Being Treated With 5-azacitidine
Brief Title: FLT-PET Imaging for MDS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HO10417; A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2012-00362 (Registry Identifier: NCI Trial ID); 2011-0285 (Other: Institutional Review Board)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-04

CONDITIONS: AML; MDS
Keywords: MDS; AML; 5 azacitidine; FLT PET

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F-FLT PET scan, 5-azacitidine treatment (Experimental): F-FLT Pet scan followed by 5-azacitidine treatment followed by FLT-PET scan. Three additional cycles of 5-azacytidine and follow up FLT-PET scan.
  Interventions: Procedure: FLT-PET scans

INTERVENTIONS:
Procedure: FLT-PET scans — FLT-PET scans prior to treatment, after Cycle 1, after Cycle 4

SUMMARY:
The main purpose of this study is to see if this tracer can be used to determine how well chemotherapy is working in patients with certain types of leukemia.

DETAILED DESCRIPTION:
Primary objectives

1. To evaluate if FLT-PET uptake shows variation during the treatment course in subjects with MDS being treated with 5-azacitidine therapy

   Secondary objectives
2. To assess FLT-PET uptake heterogeneity within given subjects being treated with 5-azacitidine therapy
3. To generate preliminary data regarding correlation between FLT-PET imaging parameters and clinical responses based on bone marrow aspirate/biopsy

ELIGIBILITY:
Inclusion Criteria:

* All subjects with previously untreated, Intermediate-2 or High risk myelodysplastic syndrome are eligible. These patients have an international prognostic scoring system (IPSS) score of 1.5 to 3.5 based on bone marrow blast percentage, karyotype, and the number of cytopenias 26.
* Subjects will receive the standard FDA-approved dose and schedule of 5-azacitidine. This dose is 75mg/m2 SQ or IV daily for seven days with cycles repeated every 28 days
* The subject's treating physician must have an initial intent of treating with at least four cycles of therapy
* Subjects must have an ECOG performance status of 0, 1, or 2
* Subjects must not have been treated with chemotherapy or radiation for another malignancy within the preceding 6 months
* Subjects must be > 18 years of age
* Subjects must have a serum creatinine < 2.0 mg/dL and/or calculated GHF 50 ml/min/1.73m (MRDR formula) or greater
* Subjects must have a serum direct bilirubin < 2.0 mg/dL unless related to Gilbert's syndrome of hemolysis. Alkaline phosphatase, SGOT (AST), and SGPT (ALT) must be less than 4 x upper limit of normal
* Women must not be pregnant nor breastfeeding
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception

Exclusion Criteria:

* Subjects who are pregnant or breast feeding
* Subjects for whom a therapy other than 5-azacitidine is recommended as first line treatment.

  * Allogeneic stem cell transplantation in patients with a suitable donor, lack of comorbidities, and good performance status

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
feasibility of using FLT-PET to assess chemotherapy response in AML/MDS | 3 years
  This pilot study is intended to investigate the feasibility of FLT-PET for early assessment of treatment response in myelodysplastic syndrome and the use of a PET isotope, (18)F-FLT, in the imaging of bone marrow in subjects with MDS. The objectives will help gather initial information for a future, larger, more definitive study.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Mattison, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States